CLINICAL TRIAL: NCT05538546
Title: The Value of Baveno VI Criteria for Screening and Monitoring of Varices Needing Treatment in Patients With Compensated Cirrhosis
Brief Title: Baveno VI Criteria in Dynamic Monitoring of High-risk Varices in Compensated Cirrhotic Patients
Acronym: CHESS2204
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Fifth Hospital of Shijiazhuang City (Other); The Sixth Hospital of Qingdao (Unknown); The Sixth Hospital of Dalian (Unknown); The Third People's Hospital of Taiyuan (Other); The Fourth People's Hospital of Qinghai Province (Other); Affiliated Hospital of Nanjing University of Chinese Medicine (Other); The Fifth People's Hospital of Wuxi Affiliated Hospital of Jiangnan University (Unknown); Beilun Hospital of Chinese Medicine (Unknown); Gansu Wuwei Tumor Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); The Third People's Hospital of Linfen City (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other); The Third Affiliated Hospital of Hebei Medical University (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Liuzhou Workers' Hospital (Other Government); The First People's Hospital of Taicang (Unknown); Xinjiang Hospital of Chinese Medicine (Unknown); Taizhou People's Hospital (Unknown); Shenzhen Third People's Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Professor, Huashan Hospital
Other Study IDs: OASIS-CHESS
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Cirrhosis; Varices; Non-invasive Evaluation
MeSH Terms: conditions — Fibrosis; Varicose Veins | interventions — Blood Cell Count; Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Population: Patients meet Baveno VI criteria (with a liver stiffness <20kPa and with a platelet count >150,000) at baseline.
  Interventions: Diagnostic Test: Complete blood count; Diagnostic Test: Transient elastrography; Diagnostic Test: Endoscopy
- Cohort 2: Population: Patients don't meet Baveno VI criteria (with a liver stiffness ≥ 20kPa or with a platelet count ≤150,000) at baseline, but don't have varices requiring treatment (proved by endoscopy at baseline)
  Interventions: Diagnostic Test: Complete blood count; Diagnostic Test: Transient elastrography; Diagnostic Test: Endoscopy

INTERVENTIONS:
Diagnostic Test: Complete blood count — Complete blood count will be conducted at 12th month and 24th month from baseline.
Diagnostic Test: Transient elastrography — Transient elastrography, and endoscopy will be conducted at 12th month and 24th month from baseline.
Diagnostic Test: Endoscopy — Endoscopy will be conducted at 12th month and 24th month from baseline.

SUMMARY:
Patients meet Baveno VI criteria (with a liver stiffness <20kPa and with a platelet count >150,000 are considered to have very low risk of having varices requiring treatment, but whether these patients can be followed up by repetition of this criteria lacks sufficient evidence. This study aimed to assess the value of Baveno VI criteria for following up and monitoring of varices needing treatment in patients with compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with liver cirrhosis diagnosed according to clinical or pathological criteria;
2. No decompensation events in the past, no ascites shown by ultrasound, no significant abnormality in liver function and coagulation function;
3. Willing to carry out routine diagnosis and treatment evaluation and follow-up liver stiffness test and gastroscopy;
4. Patients meet Baveno VI criteria (with a liver stiffness <20kPa and with a platelet count >150,000) at baseline, or patients don't meet Baveno VI criteria (with a liver stiffness ≥ 20kPa or with a platelet count ≤150,000) at baseline, but don't have varices requiring treatment (proved by endoscopy).
5. Voluntarily signed the informed consent.

Exclusion Criteria:

1. Patients with liver carcinoma;
2. Patients with portal vein thrombosis;
3. Patients with varices requiring treatment confirmed by gastroscopy during the screening period;
4. Patients who have received propranolol, ligation, sclerosis, splenectomy, transcatheter splenic arterial embolization, transjugular interhepatic portosystemicstent-shunt and other treatments to decrease portal hypertension in the past.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aimed to assess the value of Baveno VI criteria for following up and monitoring of varices needing treatment in patients with compensated cirrhosis. The study population will be patients with compensated cirrhosis, and either meet Baveno VI criteria at baseline, ordon't meet Baveno VI criteria but don't have varices requiring treatment (proved by endoscopy).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The missing rate of Baveno criteria at 12th month follow-up visit | 12 months from baseline
  The number of patients with varices requiring treatment under endoscopy divided by the number of patients meet Baveno criteria at 12th month follow-up visit

SECONDARY OUTCOMES:
The missing rate of Baveno criteria at 24th month follow-up visit | 24 months from baseline
  The number of patients with varices requiring treatment under endoscopy divided by the number of patients meet Baveno criteria at 24th month follow-up visit
Cumulative rate of decompensation events | 24 months from baseline
  The cumulative rate of decompensated events in all participants during the 24 months.
Cumulative rate of gastrointestinal bleeding | 24 months from baseline
  The cumulative rate of gastrointestinal bleeding in all participants during the 24 months.
Cumulative rate of 6-week death post gastrointestinal bleeding | 24 months from baseline
  The cumulative rate of death in 6 weeks post gastrointestinal bleeding in patients with gastrointestinal bleeding events during the 24 months.